CLINICAL TRIAL: NCT06139939
Title: Evaluation of Double Layer Graft Technique for Horizontal Ridge Augmentation With Staged Implant Placement (A Randomized Controlled Clinical Trial With Histological Assessment)
Brief Title: Guided Bone Regeneration for Horizontal Alveolar Ridge Augmentation With Double Layer Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Leila Elraee Ibrahim, assistant lecture, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Guided Bone Regeneration
Keywords: sausage technique

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- double layer technique (Experimental): include 9 patients will receive lateral alveolar ridge augmentation with double bone graft layer technique for GBR (first layer autograft followed by xenograft second layer
  Interventions: Procedure: Double layer technique
- control (Other): include 9 patients will receive lateral alveolar ridge augmentation with stander protocol for GBR technique (mixture of autograft and xenograft
  Interventions: Procedure: Double layer technique

INTERVENTIONS:
Procedure: Double layer technique — Double layer technique for alveolar ridge augmentation (first layer autograft followed by xenograft second layer).

SUMMARY:
clinical study with guided bone regeneration for deficient alveolar ridge to restore the defect in width and be able to place implant with two different technique

DETAILED DESCRIPTION:
This study will be conducted to compare the bone formation with double layer graft technique versus standard protocol in GBR for horizontal ridge augmentation with staged implant placement

Primary outcome: Evaluation of alveolar bone width gain clinically and radiographically.

Secondary outcome: Histological analysis of remodeled bone.

ELIGIBILITY:
Inclusion Criteria:

* 1- Healthy adult patients as evidenced by Burkett's oral medicine health history questionnaire. (American Society of Anesthesiologists I; ASA I) (Mombelli and Cionca, 2006) 2- Both genders. 3- Age from 20 - 40 years old. 4- Having missing maxillary or mandibular tooth with low or moderate horizontal defect (4-8) according to cologne classification (2013) 5- Presence of sufficient bone height minimum 12 mm that does not require bone grafting or any other ridge augmentation procedure.(Shah and Lum, 2008) 6- Presence of sufficient keratinized mucosa of at least 2 mm.(Bassetti, et al. 2015)

Exclusion Criteria:

* 1- Smokers (Twito and Sade, 2014) 2- Vulnerable groups (as pregnant females and decisional impaired individuals) will be excluded from the study.

  3- Patients with poor oral hygiene or not willing to perform oral hygiene measures.

  4- Prisoners and handicapped patients. 5- Patients with periodontal or periapical infections.(Tonetti, et al. 1996)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
clinical and radiographic outcome | 6 months
  clinical ridge width gain

SECONDARY OUTCOMES:
histological analysis of remodeled bone. | 6 months
  core biopsy were taken after 6 months from augmentation

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university , faculty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided